CLINICAL TRIAL: NCT02632383
Title: Young With Diabetes Type 1 - Test of an mHealth App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Herlev Hospital (Other); Steno Diabetes Center Copenhagen (Other); Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2015-12-02; First posted 2015-12-16 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes type 1; Transition; Telemedicine; mHealth app; Youth; Self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental): Intervention: Young with Diabetes - app The test group receives standard care and the mHealth app "Young with Diabetes" - app to support young people to self-manage their diabetes.
  The young people's parents are also invited to download the app. The diabetes team (doctors, nurses and dieticians) also have the app and uses the app in their consultations with the young people.
  Interventions: Device: Young with Diabetes - app
- Control Group (No Intervention): The control group receives standard care

INTERVENTIONS:
Device: Young with Diabetes - app — The mHealth app "Young with Diabetes" containes 8 main functions:
  1. Contact your health care provider (ask questions, set the agenda for the next clinical visit)
  2. My Department (hotline numbers, videos about the new adult department, pictures of my diabetes team)
  3. Chatroom
  4. Counting Carbohydrates (information and tips about carbs, introduction to apps to count carbs, quiz)
  5. Knowledge-section (Text, links, tips and videos (animations and videoselfies) about What is diabetes?, Alcohol etc.)
  6. Tips packages (Receive a tip about alcohol, drivers license etc.)
  7. To parents (Text, links, tips and videoselfies to parents about what it is like to be young with diabetes and what they can do to support)
  8. Reminder
  Arms: Test Group

SUMMARY:
A multicenter randomized controlled trial testing the app "Young with Diabetes"

DETAILED DESCRIPTION:
Young people with diabetes type 1, their parents and health care providers have participated in developing the mHealth app "Young with Diabetes".

The aim of the app is to support young people to self-manage their diabetes type 1.

A test group of 70 young people with diabetes type 1 test the app for 12 months as a supplement to standard care and the control group receives standard care only.

At baseline and after 2, 7 and 12 months HbA1c, problem areas in diabetes, perceived competences in diabetes and health care climate are measured.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* 14 to 22 years old
* followed at one of the six diabetes departments/centers

  1. Pediatric and Adolescent Department, Nordsjællands Hospital, Hillerød
  2. Department of Cardiology, Nephrology and Endocrinology, Nordsjællands Hospital, Hillerød
  3. Pediatric and Adolescent Department, Herlev Hospital
  4. Steno Diabetes Center, Gentofte
  5. Pediatric Department, Roskilde Hospital
  6. Department of Endocrinology, Køge Hospital
* have an iOS or android smartphone
* last measured HbA1c before sending out recruiting letters: 64 mmol/mol or more (if the last measured HbA1c is older than 6 months at time of baseline visit a new HbA1c is measured and has to be at least 64 mmol/mol before the participant kan be randomized)
* mean of the three last measured HbA1c before sending out recruiting letters: 58 mmol/mol or more (if the third last HbA1c is older than 18 months at time of baseline visit a new HbA1c is measured and has to be at least 64 mmol/mol before the participant kan be randomized)

Exclusion Criteria:

* A psychical or psychiatric disorder that enables them to use the app
* Participates in other diabetes interventions
* Sees a psychologist or psychiatrist
* Have participated in developing the app Young with Diabetes

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Glycemic control measured by HbA1c | Glycemic control is measured by HbA1c at 12 months

SECONDARY OUTCOMES:
Problem areas in diabetes measured by PAID-20 | Problem areas in diabetes are measured by PAID-20 at 12 months
Perceived competences in diabetes measured by PCD-questionnaire | Perceived competences in diabetes are measured by PCD-questionnaire at 12 months
Health Care Climate measured by HCCQ-questionnaire | Health Care Climate is measured by HCCQ-questionnaire at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Castensøe-Seidenfaden, Principal Investigator — Pediatric and Adolescent Department, Nordsjællands Hospital, Hillerød
Locations (6):
- Denmark (6):
  - Steno Diabetes Center, Gentofte Municipality, Gentofte
  - Pediatric and Adolescent Department, Herlev Hospital, Herlev, Herlev
  - Department of Cardiology, Nephrology and Endocrinology, Nordsjællands Hospital, Hillerød, Hillerød, Hillerød
  - Pediatric and Adolescent Department, Nordsjællands Hospital, Hillerød, Hillerød, Hillerød
  - Department of Endocrinology, Køge Hospital, Køge, Køge
  - Pediatric Department, Roskilde Hospital, Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castensoe-Seidenfaden P, Husted GR, Jensen AK, Hommel E, Olsen B, Pedersen-Bjergaard U, Kensing F, Teilmann G. Testing a Smartphone App (Young with Diabetes) to Improve Self-Management of Diabetes Over 12 Months: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jun 26;6(6):e141. doi: 10.2196/mhealth.9487. PMID 29945861